CLINICAL TRIAL: NCT04306237
Title: A Randomized, Double-Blinded, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Efficacy of IMB-1018972 in Patients With Refractory Angina
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of IMB-1018972 in Patients With Refractory Angina
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Coronavirus pandemic
Sponsor: Imbria Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIMB-8972-201
Record Dates: First submitted 2020-03-08; First posted 2020-03-12 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Refractory Angina
MeSH Terms: conditions — Angina Pectoris

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IMB-1018972 (Experimental): Participants will receive IMB-1018972 (200 mg) MR tablets twice daily for 16 weeks
  Interventions: Drug: IMB-1018972
- Placebo (Placebo Comparator): Participants will receive matching placebo tablets twice daily for 16 weeks
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: IMB-1018972 — IMB-1018972 200 mg tablet for oral administration
  Arms: IMB-1018972
Drug: Placebo oral tablet — Matched placebo tablet for oral administration
  Arms: Placebo

SUMMARY:
The objectives of the study are to assess the safety, tolerability, and potential efficacy of IMB-1018972 on patients with refractory angina. Study will assess functional capacity employing a modified Bruce Protocol treadmill ETT, patient reports of angina symptoms via an electronic diary, and activity using an accelerometer.

ELIGIBILITY:
Inclusion Criteria:

1. Is between the ages of 18 and 85 years, inclusive.
2. Is capable of understanding the written informed consent, and providing signed, dated, and witnessed written informed consent.
3. Has complied with and is willing to continue to comply with the specified procedures (eg, angina diary during screening) and complete specific follow-up evaluations.
4. Has coronary artery disease confirmed by at least one of the following:

   * Documented prior MI, CABG surgery, or PCI -OR-
   * Angiography performed within the 24 months prior to Visit 1 confirming CAD (eg, evidence of ≥70% stenosis of at least one major coronary artery or diffuse CAD).
5. Has evidence of stress induced ischemia documented by either:

   * Protocol-specified ETT ECG demonstrating at least 0.5 mm exercise-induced ST segment depression with onset <9 minutes on at least 1 of the screening ETTs -OR-
   * Prior evidence of stress-induced reversible perfusion defect in the last 24 months (without intervening revascularization) identified by at least one of the following:

     * Radionuclide imaging study
     * Echocardiographic imaging study
     * FFR <0.8
     * IFR <0.89
     * FFR CT <0.8
     * CFR <2.5
6. Has a minimum 3 month history of exertional angina, including angina with a minimum frequency of 2 anginal episodes per week on average for the 2 weeks prior to enrolling in the study while on optimal guideline directed medical therapy for their angina.
7. Is on optimal, dual agent, antianginal therapy for their angina for at least 1 month prior to the first screening ETT. Consistent with ACC/AHA and ESC Class I guideline directed medical therapy (GDMT), criteria for optimal therapy include treatment with both: (a) a beta-adrenergic blocking agent and treatment with (b) a calcium channel blocker OR a long-acting nitrate. If unacceptable side effects are intolerable and documented with a therapy listed in (a) or (b), treatment with only 1 antianginal medication is acceptable. Additionally, patients should be treated with short-acting nitrates per GDMT.
8. Is currently not clinically indicated for coronary revascularization (ie, PCI or CABG) in the opinion of the principle investigator at the time of screening through 6 months after randomization.
9. Has a CCS score of II, III or stabilized IV for 1 month prior to screening.
10. Meets the following requirements after 2 screening modified Bruce protocol ETTs:

    a. Stopping the treadmill test due to angina on each test b. Total exercise duration must fall between 3 and 9 minutes on each test c. To document inducible myocardial ischemia: i. For those patients with interpretable ECGs, at least 0.5 mm exercise induced ST segment depression must occur with onset <9 minutes on at least 1 of the screening ETTs.

    d. Difference in TED between the 2 qualifying ETTs must not exceed 20% of the longer test or 1 minute, whichever limit is smaller.

    e. Consideration of a third ETT may be discussed by the investigator with the study medical monitor, who may authorize the performance of a third ETT a minimum of 5 days and no more than 10 days after the second ETT

Exclusion Criteria:

1. If any of the following have occurred:

   * Use of TMZ anytime in prior history
   * In the prior 6 months:

     * Diagnosis of NYHA Class 3 or 4 (heart failure)
     * Hospitalization for heart failure
     * Coronary artery bypass graft surgery
     * Cardiac resynchronization therapy placement or adjustments to CRT parameters
     * Implantable cardioverter defibrillator or biventricular pacemaker placement
   * In the prior 3 months:

     * Hospitalization for a cardiovascular indication
     * Cerebral vascular accident
     * Transient ischemic attack
     * Percutaneous coronary intervention
   * In the prior 1 month:

     * Use of perhexiline or meldonium.
2. Has a history of moderate to severe valvular heart disease defined as aortic stenosis (valve area <1.5 cm2), aortic insufficiency, mitral stenosis (valve area <1.5 cm2), or mitral valve regurgitation of grade 3 or worse.
3. Has significant hepatic disease, with increased liver function tests such as total bilirubin, aspartate aminotransferase, or alanine aminotransferase more than 2 times of ULN at baseline (excluding patients with documented history of Gilbert syndrome).
4. Has severe renal impairment (ie, creatinine clearance <30 mL/min at screening, measured using 4-variable modification of diet in renal disease equation).
5. Has a history of Parkinson disease, Parkinsonian symptoms, tremors, restless leg syndrome, or other related movement disorders.
6. Has a history of vasospastic angina or microvascular angina.
7. Has an exacerbating cause for angina (eg, anemia [ie, hemoglobin <10 g/dL], uncontrolled hypertension [ie, BP ≥160/90 mmHg], hyperthyroid, or rapid AF [ie, AF with average rate >120 beats per minute]) at screening.
8. Has long-QT and life-threatening LV arrhythmia.
9. Has comorbidities limiting life expectancy to less than 3 years.
10. Is pregnant, planning pregnancy, or lactating.
11. Has a history of alcohol abuse or drug addiction.
12. Has a positive test for drugs (eg, opiates, methadone, cocaine, amphetamines [including ecstasy], or barbiturates) at screening.
13. Has a positive test for HBsAg, HCV antibodies, or HIV1/2 antibodies at screening.
14. Is participating in another research study.
15. Is an employee or family member of the investigator or study site personnel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Modified Bruce Protocol Treadmill ETT | 8 weeks
  Change from baseline to Week 8 in total exercise duration (seconds)
Safety and Tolerability of IMB-1018972 in Patients with Refractory Angina | 16 weeks
  Incidence of AEs, changes from baseline in physical examinations, vital signs, clinical laboratories, and ECG

SECONDARY OUTCOMES:
Assess the benefit of IMB-1018972 on patient report of angina symptoms employing an electronic diary | 16 weeks
  Change from baseline per week in the incidence of angina symptoms
Assess the potential treatment benefit of IMB-1018972 on patient report of rescue NTG use employing an electronic diary | 16 weeks
  Change from baseline in daily counts of NTG use
Assess the potential treatment benefit of IMB-1018972 on patient activity employing a wearable device | 16 weeks
  Change from baseline in total daily activity at Week 16 (activity units)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Chamberlin, MD, Study Director — Imbria Pharmaceuticals
Locations (1):
- Imbria Investigational Site, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No